CLINICAL TRIAL: NCT00964795
Title: An Open-label, Long-term, Safety and Tolerability Extension Study of Intravitreal VEGF Trap-Eye in Neovascular Age-Related Macular Degeneration
Brief Title: Open-label Extension Study of Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) in Neovascular ("Wet") Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFT-OD-0910
Record Dates: First submitted 2009-08-20; First posted 2009-08-25 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Eyes; Neovascular; Macular Degeneration; Retina; AMD; VEGF Trap-Eye; Best Corrected Visual Acuity
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label Intravitreal Aflibercept Injection (Experimental): Open-label Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) 2mg (40 mg/mL) was administered no more frequently than every 4 weeks, but no less frequently than every 12 weeks until amendment 4. Starting with amendment 4, Intravitreal Aflibercept Injection was administered no less frequently than every 8 weeks. Within these limits, the investigator would determine the interval of Intravitreal Aflibercept Injection administration on an as-needed basis according to the protocol-suggested re-treatment criteria, however the injections must have occurred at least every 12 weeks prior to amendment 4, and at least every 8 weeks starting from amendment 4 as noted above.
  Interventions: Drug: Intravitreal Aflibercept Injection 2mg

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection 2mg
  Other Names: IAI; EYLEA®; BAY86-5321; VEGF Trap-Eye

SUMMARY:
The primary objective is to assess long-term safety and tolerability of Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) in patients with neovascular AMD.

DETAILED DESCRIPTION:
The dose evaluated in this study, Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) 2mg, will be the higher of the 2 dose strengths evaluated in parent study VGFT-OD-0605 (NCT00509795) and is the dose level administered in study VGFT-OD-0702 (NCT00527423), a long-term open-label extension study. For these reasons, this dose has been selected for this extension study.

Participants will be seen in the clinic for quarterly visits starting with day 1 to assess safety. Study drug will be administered on an as-needed basis at the discretion of the investigator with a minimum allowed interval of every 4 weeks and a maximum allowed interval of every 12 weeks. This study will assess the frequency that re-treatment is needed and the effect of continued Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) treatment on BCVA.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Study VGFT-OD-0605 through week 96.
* In the opinion of the investigator, the study eye has neovascular AMD and may continue to require treatment.

Exclusion Criteria:

* Presence of any condition that would jeopardize the patient's participation in this study.
* Females who are pregnant, breastfeeding, or of childbearing potential, unwilling to practice adequate contraception throughout the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2009-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (124):
- United States (115):
  - Birmingham (2 Locations), Alabama
  - Phoenix (2 Locations), Arizona
  - Tucson (2 Locations), Arizona
  - Arcadia, California
  - Beverly Hills, California
  - Campbell, California
  - Fresno, California
  - Fullerton, California
  - La Jolla, California
  - Loma Linda, California
  - Mountain View, California
  - Oakland, California
  - Orange, California
  - Palm Desert, California
  - Sacramento, California
  - San Mateo, California
  - Santa Ana, California
  - Torrance, California
  - Westlake Village, California
  - Yorba Linda, California
  - Colorado Springs, Colorado
  - Denver (2 Locations), Colorado
  - Bridgeport, Connecticut
  - New Haven, Connecticut
  - New London, Connecticut
  - Altamonte Springs, Florida
  - Boynton Beach, Florida
  - Fort Myers (2 Locations), Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando (2 Locations), Florida
  - Oscala, Florida
  - Palm Beach Gardens, Florida
  - Pensacola, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - ‘Aiea, Hawaii
  - Glenview, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - New Albany, Indiana
  - Iowa City, Iowa
  - Wichita, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Bangor, Maine
  - Portland, Maine
  - Baltimore (3 Locations), Maryland
  - Chevy Chase, Maryland
  - Hagerstown, Maryland
  - Boston (2 Locations), Massachusetts
  - Peabody, Massachusetts
  - Ann Arbor, Michigan
  - Battle Creek, Michigan
  - Grand Rapids, Michigan
  - Jackson, Michigan
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Florissant, Missouri
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Portsmouth, New Hampshire
  - Lawrenceville, New Jersey
  - Northfield, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Lynbrook, New York
  - New York (6 Locations), New York
  - Rochester (2 Locations), New York
  - Slingerlands, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Ashland, Oregon
  - Portland (3 Locations), Oregon
  - Salem, Oregon
  - Kingston, Pennsylvania
  - Philadelphia (3 Locations), Pennsylvania
  - Pittsburgh (2 Locations), Pennsylvania
  - West Mifflin, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Austin (3 Locations), Texas
  - Dallas, Texas
  - Fort Worth (2 Locations), Texas
  - Houston, Texas
  - McAllen, Texas
  - Odessa, Texas
  - San Antonio (2 Locations), Texas
  - Tyler, Texas
  - Salt Lake City (2 Locations), Utah
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison (2 Locations), Wisconsin
  - Milwaukee, Wisconsin
- Canada (9):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Montreal (2 Locations), Quebec
  - Regina, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After informed consent was obtained, the 323 participants who completed the parent study, VGFT-OD-0605 (NCT00509795), and met the protocol eligibility criteria, were enrolled at 71 clinical sites in the US & Canada. The first visit occurred concurrently with the last visit in the parent study. The last participant entered this study on 18-May-2011.
Pre-assignment Details: Intravitreal Aflibercept Injection [commercially known EYLEA® (aflibercept) Injection] was approved in the US for treatment of neovascular ("wet") age-related macular degeneration (AMD) as the study was ongoing. For collection of long-term safety and best corrected visual acuity data on EYLEA®, the study was extended in the US from 30 to 45 months.
Period: Overall Study
Arm/Group | Open-label Intravitreal Aflibercept Injection
Started | 323 (randomized)
Number of Participants Treated | 320
Completed | 16 (Prior to amendment 4, 16 participants completed up to Week 120. No participants completed Week 180.)
Not Completed | 307
Not completed — Withdrawal by Subject | 79
Not completed — Adverse Event | 12
Not completed — Death | 14
Not completed — Lost to Follow-up | 7
Not completed — Termination of Study by Sponsor | 169
Not completed — Unwilling to sign ICF for amendment 4 | 3
Not completed — Other | 23

BASELINE CHARACTERISTICS:
Population: Randomized participants included all participants who were enrolled in the study. The data were used to analyze the safety and efficacy parameters to characterize the long-term effect of Intravitreal Aflibercept Injection treatment. The average study duration for all enrolled participants was 116.9 weeks.
Arm/Group | Open-label Intravitreal Aflibercept Injection
Number analyzed (Participants) | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 127

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Intravitreal Aflibercept Injection in Participants With Neovascular AMD
Description: The primary endpoint in the study is the safety and tolerability of Intravitreal Aflibercept Injection in patients with neovascular AMD (Age-related Macular Degeneration) from day 1 through the end of treatment visit (week 180) based on the number of participants who experienced any treatment-emergent adverse event (TEAE).
  Treatment-emergent adverse events were categorized according to Ocular TEAEs in the study eye, Ocular TEAEs in the fellow eye, and Non-Ocular TEAEs
Time Frame: Baseline (day 1) through end of treatment (Week 180)
Measure: Number; unit: participants
Groups:
- Open-label Intravitreal Aflibercept Injection: Open-label Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) 2 mg (40 mg/mL) was administered no more frequently than every 4 weeks, but no less frequently than every 12 weeks until amendment 4. Starting with amendment 4, Intravitreal Aflibercept Injection was administered no less frequently than every 8 weeks. Within these limits, the investigator would determine the interval of Intravitreal Aflibercept Injection administration on an as-needed basis according to the protocol-suggested re-treatment criteria, however the injections must have occurred at least every 12 weeks prior to amendment 4, and at least every 8 weeks starting from amendment 4 as noted above.
Arm/Group | Open-label Intravitreal Aflibercept Injection
Number analyzed (Participants) | 323
participants
  Number of participants with any TEAE | 290
  Any ocular TEAE | 239
  Any ocular TEAE: Study eye | 204
  Any ocular TEAE: Fellow eye | 169
  Any non-ocular TEAE | 232
  Any serious TEAE | 105
  Discontinuation of study due to AE | 12
  Any Death due to TEAE | 17

2. Secondary Outcome: Change in BCVA Letter Score (mLOCF)
Description: The secondary endpoint in the study is the change in BCVA letter score from baseline through Week 116.
  (mLOCF: The last non-missing observation prior to the missing visit was carried forward to impute the missing data; no imputation after last visit; no baseline value carried forward).
Time Frame: Baseline through Week 116
Measure: Mean (Standard Deviation); unit: letters correctly read
Arm/Group | Open-label Intravitreal Aflibercept Injection
Number analyzed (Participants) | 323
letters correctly read | -2.7 (12.50)

3. Other Pre Specified Outcome: Summary of Treatment Duration (Weeks)
Description: Treatment Duration = (last dose date - first dose date + 28)/7
Time Frame: Baseline through end of treatment (Week 180)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Open-label Intravitreal Aflibercept Injection
Number analyzed (Participants) | 323
weeks | 110.4 (42.16)

4. Other Pre Specified Outcome: Summary of Study Duration (Weeks)
Description: Study Duration = (last visit/ discontinuation date - first dose date + 28)/7
Time Frame: Baseline through end of treatment (Week 180)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Open-label Intravitreal Aflibercept Injection
Number analyzed (Participants) | 323
weeks | 116.9 (44.3)

ADVERSE EVENTS:
Groups:
- Open-label Intravitreal Aflibercept Injection: Open-label Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) 2 mg (40 mg/mL) was administered no more frequently than every 4 weeks, but no less frequently than every 12 weeks until amendment 4. Starting from amendment 4, Intravitreal Aflibercept Injection was administered no less frequently than every 8 weeks. Within these limits, the investigator would determine the interval of Intravitreal Aflibercept Injection administration on an as-needed basis according to the protocol-suggested re-treatment criteria, however the injections must have occurred at least every 12 weeks prior to amendment 4, and at least every 8 weeks starting from amendment 4 as noted above.
Arm/Group | Open-label Intravitreal Aflibercept Injection
Serious Adverse Events (participants affected / at risk) | 105/323
Other Adverse Events (participants affected / at risk) | 102/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Intravitreal Aflibercept Injection (N=323)
Anaemia (Blood and lymphatic system disorders) | 2
Coagulopathy (Blood and lymphatic system disorders) | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 5
Angina Pectoris (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 12
Bundle Branch Block Right (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 4
Cardiac Failure Acute (Cardiac disorders) | 3
Cardiac Failure Congestive (Cardiac disorders) | 3
Cardiogenic Shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 4
Myocardial Infarction (Cardiac disorders) | 4
Myocardial Rupture (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Appendix Disorder (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis Ischaemic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal Angiodysplasia Haemorrhagic (Gastrointestinal disorders) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 1
Device Dislocation (General disorders) | 1
Multi-Organ Failure (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Biliary Dyskinesia (Hepatobiliary disorders) | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1
Hepatic Haemorrhage (Hepatobiliary disorders) | 1
Anaphylactic Reaction (Immune system disorders) | 1
Abdominal Abscess (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchitis Viral (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Clostridium Difficile Colitis (Infections and infestations) | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis Norovirus (Infections and infestations) | 1
Gastroenteritis Viral (Infections and infestations) | 1
Pericolic Abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia Bacterial (Infections and infestations) | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1
Pneumonia Viral (Infections and infestations) | 1
Pyelonephritis Acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Septic Shock (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 5
Urosepsis (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 2
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 16
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 2
Humerus Fracture (Injury, poisoning and procedural complications) | 3
Pancreatic Leak (Injury, poisoning and procedural complications) | 1
Radius Fracture (Injury, poisoning and procedural complications) | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1
Splenic Rupture (Injury, poisoning and procedural complications) | 2
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 1
Blood Pressure Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Bone Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid Artery Stenosis (Nervous system disorders) | 1
Cerebral Haemorrhage (Nervous system disorders) | 1
Cerebral Infarction (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 5
Convulsion (Nervous system disorders) | 1
Embolic Stroke (Nervous system disorders) | 1
Facial Neuralgia (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Hypertensive Encephalopathy (Nervous system disorders) | 1
Intracranial Haematoma (Nervous system disorders) | 1
Ischaemic Stroke (Nervous system disorders) | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 8
Transient Ischaemic Attack (Nervous system disorders) | 4
Major Depression (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 3
Psychotic Disorder (Psychiatric disorders) | 1
Calculus Ureteric (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Obstructive Uropathy (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 4
Renal Failure Chronic (Renal and urinary disorders) | 1
Ureteric Obstruction (Renal and urinary disorders) | 1
Uterine Polyp (Reproductive system and breast disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1
Perivascular Dermatitis (Skin and subcutaneous tissue disorders) | 1
Colectomy (Surgical and medical procedures) | 1
Medical Device Removal (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Retinal Haemorrhage (Eye disorders) | 1
Angle Closure Glaucoma (Eye disorders) | 1 — Study eye
Cataract (Eye disorders) | 1 — Study eye
Glaucoma (Eye disorders) | 1 — Study eye
Retinal Haemorrhage (Eye disorders) | 2 — Study eye
Retinal Oedema (Eye disorders) | 1 — Study eye
Visual Acuity Reduced (Eye disorders) | 1 — Study eye
Device Dislocation (General disorders) | 1 — Study eye
Endophthalmitis (Infections and infestations) | 3 — Study eye
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 — Study eye
Intraocular Pressure Increased (Investigations) | 1 — Study eye
Femur Fracture (Injury, poisoning and procedural complications) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Intravitreal Aflibercept Injection (N=323)
Nausea (Gastrointestinal disorders) | 22
Bronchitis (Infections and infestations) | 19
Nasopharyngitis (Infections and infestations) | 22
Upper Respiratory Tract Infection (Infections and infestations) | 20
Fall (Injury, poisoning and procedural complications) | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 17
Hypertension (Vascular disorders) | 29
Age-Related Macular Degeneration (Eye disorders) | 30
Retinal Haemorrhage (Eye disorders) | 39
Cataract (Eye disorders) | 17 — Study eye
Conjunctival Haemorrhage (Eye disorders) | 30 — Study eye
Posterior Capsule Opacification (Eye disorders) | 18 — Study eye
Retinal Detachment (Eye disorders) | 17 — Study eye
Retinal Haemorrhage (Eye disorders) | 34 — Study eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator (PI) may publish results provided a copy of oral/ written publication is received by sponsor at least 45 days in advance for review & comment. If the parties disagree, PI agrees to meet with sponsor prior to submission to resolve any disagreement. Sponsor reserves the right to remove confidential information from such submission. It is also agreed that publication of results shall be made only as part of a publication of the results obtained by all sites performing the study.